CLINICAL TRIAL: NCT01974765
Title: A Phase II Trial of Enzalutamide in Patients With Androgen Receptor Positive (AR+) Ovarian, Primary Peritoneal or Fallopian Tube Cancer and One, Two or Three Prior Therapies
Brief Title: Enzalutamide in Patients With Androgen Receptor Positive (AR+) Ovarian, Primary Peritoneal or Fallopian Tube Cancer and One, Two or Three Prior Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-119
Record Dates: First submitted 2013-10-25; First posted 2013-11-04 (Estimated); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-03

CONDITIONS: Advanced Epithelial Ovarian; Recurrent Epithelial Ovarian; Fallopian Tube; Primary Peritoneal Carcinoma
Keywords: Enzalutamide; Androgen Receptor Positive (AR+); 13-119
MeSH Terms: interventions — enzalutamide

ARMS (1):
- Enzalutamide (Experimental): After signing a screening consent, patients archival tissue will be evaluated for degree of AR positivity by AR staining. Patients with no archival tissue available will undergo a biopsy (using the modality deemed most appropriate by the patient's physician) for collection of tumor tissue for AR positivity by IHC. Only AR+ patients, defined as ≥5 % positivity by IHC, will be included. All IHC testing will be performed in the MSKCC Clinical CLIA approved laboratory.
  All enrolled patients will be treated with enzalutamide 160 mg by mouth QD until progression of disease (POD), unacceptable toxicity or withdrawal from study. All treatments will be administered in the outpatient setting.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — All enrolled patients will be treated with enzalutamide 160mg by mouth QD. Study drugs will be self-administered by patients. A cycle is 28 days.

SUMMARY:
This is a Phase II study. The purpose of this study is to find out what effects, good and/or bad enzalutamide has on the patient and the cancer. All patients who enter the study will be closely monitored for side-effects. If multiple patients develop significant side effects from enzalutamide, the study may be stopped early.

Enzalutamide is an androgen-receptor inhibitor, which means that it blocks the activity of the hormone testosterone. In ovarian, fallopian tube, and primary peritoneal cancers that express the androgen receptor, blocking the androgen-receptor may possibly slow or stop tumor growth. Enzalutamide has been studied in women with breast cancer, but this is the first study using enzalutamide for the treatment of patients with ovarian, primary peritoneal, or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma. Histologic documentation of the original primary tumor is required via the pathology report
* AR expression ≥5% by IHC. In cases where multiple blocks are available staining will be performed on unstained slides from 3 separate blocks. If ≥ 5% AR tumor staining is seen on ≥ 1 slide the tumor will be considered to be AR+.
* Patients with the following histologic cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial adenocarcinoma, transitional cell carcinoma, malignant Brenner's tumor, or adenocarcinoma not otherwise specified
* Measurable disease as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension. Each lesion must be ≥10mm when measured by CT, MRI or caliper measurement by clinical exam; or ≥ 20mm when measured by chest x-ray. Lymph nodes must be ≥ 15mm in short axis when measured by CT or MRI
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease
* Patients may have received, but are not required to have received, one or two additional cytotoxic regimens for management of recurrent or persistent disease
* Patients who have received only one prior cytotoxic regimen (platinum-based regimen management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* Patients are allowed to receive, but are not required to receive, non-cytotoxic therapy (such as bevacizumab) as part of their primary treatment regimen.
* Patients are allowed to receive, but are not required to receive, non-cytotoxic therapy for management of recurrent or persistent disease
* Must be ≥ 18 years of age
* Karnofsky Performance Status (KPS) of ≥ 70%
* Life expectancy of ≥ 12 weeks Women of child-bearing potential must have a negative pregnancy test within 14 days prior to commencement of study treatment
* Women of child bearing potential must use an effective form of contraception during study and for at least 6 months after completion of study treatment
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * At least 4 weeks out from their last dose of radiation therapy
  * At least 4 weeks post-op from any major surgical procedure
  * At least 3 weeks out from their last dose of chemotherapy and/or biologic/targeted therapy
* No prior hormonal therapy for treatment of cancer within the past 21 days
* Absence of any psychological, familial, sociological or geographic condition that would potentially hamper compliance with the study protocol
* Prior use of or participation in a clinical trial evaluating and agent that either blocks androgen synthesis (e.g. abiraterone acetate, TAK-700, TAK-683, TAK-448) or targets the AR (e.g., bicalutamide, BMS-641988) (patients who are known to have only received placebo in these studies are eligible)
* Laboratory Test Findings performed within 14 days prior to initiation of study drug showing:

Bone marrow function:

Absolute neutrophil count (ANC) ≥ 1,000/mcL Platelets ≥ 100,000/mcL Hemoglobin ≥ 8 g/dL o Renal function: Creatinine ≤ 1.5 x ULN

o Hepatic function: Bilirubin ≤ 1.5 x ULN AST and ALT ≤ 2.5 x ULN

* Resolution of all acute toxic effects of prior therapy to NCI CTCAE (Version 4.0) Grade ≤ 1, with the exception of unresolved Grade 2 neuropathy and Grade 2 alopecia, which are allowed
* Patients must be able to swallow tablets whole, without crushing

Exclusion Criteria:

* A history of another invasive malignancy (other than non-melanoma skin cancer or curatively treated in situ carcinoma) with evidence of disease within the past 3 years
* Use of a medication known to lower the seizure threshold within 28 days of first dose of study drug
* Known brain metastasis
* History of seizure
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95mmHg) despite medical treatment. Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
* Clinically significant heart disease as evidenced by myocardial infarction or arterial thrombotic event within the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline
* Refractory nausea and vomiting, requirement for parenteral hydration and/or nutrition, drainage gastrostomy tube, malabsorption, external biliary shunt, or significant small bowel resection that would preclude adequate study drug absorption
* Anticipated or ongoing administration of anti-cancer therapies other than those administered in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Grisham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzalutamide: After signing a screening consent, patients archival tissue will be evaluated for degree of AR positivity by AR staining. Patients with no archival tissue available will undergo a biopsy (using the modality deemed most appropriate by the patient's physician) for collection of tumor tissue for AR positivity by IHC. Only AR+ patients, defined as ≥5 % positivity by IHC, will be included. All IHC testing will be performed in the MSKCC Clinical CLIA approved laboratory.
  All enrolled patients will be treated with enzalutamide 160 mg by mouth QD until progression of disease (POD), unacceptable toxicity or withdrawal from study. All treatments will be administered in the outpatient setting.
  Enzalutamide: All enrolled patients will be treated with enzalutamide 160mg by mouth QD. Study drugs will be self-administered by patients. A cycle is 28 days.
Period: Overall Study
Arm/Group | Enzalutamide
Started | 59
Completed | 55
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 64 [29 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 48
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Number (90% Confidence Interval); unit: percentage of participants with response
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
percentage of participants with response | 1.7 [0.2 to 100]

2. Primary Outcome: Partial Response
Description: as for outcome 1
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
Participants
  Partial Response | 1
  No Partial Response | 58

3. Secondary Outcome: Number of Participants Assessed for Treatment-Related Adverse Events
Description: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0. For each symptom i.e., frequency, severity, the worst score experienced by the patient will be recorded
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
Participants | 59

4. Secondary Outcome: Median Androgen Receptor/AR Expression Levels on Tissue
Description: Median Androgen Receptor/AR expression levels on tissue will be determined using standard immunohistochemistry methodology
Time Frame: 2 years
Measure: Median (Full Range); unit: ng/dL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
ng/dL | 60 [5 to 99]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 35/59
Serious Adverse Events (participants affected / at risk) | 9/59
Other Adverse Events (participants affected / at risk) | 14/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=59)
Abdominal infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=59)
Fatigue (General disorders) | 14
Hot flashes (Vascular disorders) | 12
Diarrhea (Gastrointestinal disorders) | 8
Hypertension (Vascular disorders) | 8
Insomnia (Psychiatric disorders) | 8
Nausea (Gastrointestinal disorders) | 8
Headache (Nervous system disorders) | 7
Abdominal Pain (Gastrointestinal disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Anemia (Blood and lymphatic system disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5
Dysgeusia (Nervous system disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Memory impairment (Nervous system disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anxiety (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Malaise (General disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Palpitations (Cardiac disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT01974765/Prot_SAP_000.pdf